CLINICAL TRIAL: NCT00654368
Title: Canadian Methotrexate and Etanercept Outcome Study: An Open Label Randomized Trial of Etanercept and Methotrexate Versus Etanercept Alone in the Treatment of Rheumatoid Arthritis (CAMEO)
Brief Title: CAMEO: Canadian Methotrexate and Etanercept Outcome Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070301
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Amgen
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etanercept + Methotrexate (Active Comparator): After six months of treatment with 50 mg/week subcutaneous etanercept added to existing methotrexate therapy of at least 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses) participants were randomized to continue both etanercept plus methotrexate for an additional 18 months.
  Interventions: Biological: Etanercept; Drug: Methotrexate
- Etanercept Only (Experimental): After six months of treatment with 50 mg/week subcutaneous etanercept added to existing methotrexate therapy of at least 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses) participants were randomized to discontinue methotrexate (tapered over 6 weeks) and continue etanercept alone for an additional 18 months.
  Interventions: Biological: Etanercept; Drug: Methotrexate

INTERVENTIONS:
Biological: Etanercept — Commercially available etanercept administered subcutaneously at 50 mg/week.
  Other Names: Enbrel®
Drug: Methotrexate — Commercially available methotrexate administed orally, subcutaneously or intramuscularly 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses)

SUMMARY:
The purpose of the study is to evaluate the use of etanercept in the treatment of rheumatoid arthritis with or without methotrexate treatment over a 24 month period

DETAILED DESCRIPTION:
This noninferiority study was a multicenter, open-label, randomized trial of patients with rheumatoid arthritis (RA). Patients who did not have an adequate response to methotrexate (MTX) had etanercept (50 mg/week subcutaneously [SC]) added to existing MTX therapy of at least 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses of MTX) at baseline and were followed for 6 months. After 6 months of therapy, participants were randomized in a 1:1 ratio to one of the 2 treatment arms: either discontinue MTX (tapered over 6 weeks) and continue etanercept alone or continue both etanercept plus MTX for an additional 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the baseline visit
* An American College of Rheumatology(ACR) diagnosis of rheumatoid arthritis with onset of symptoms of at least 6 months
* Active disease of at least 3 swollen joints from the Disease Activity Severity 28 at the baseline visit
* A Disease Activity Severity 28 score of ≥ 3.2 at the baseline visit
* Have not previously received etanercept therapy
* Able to start etanercept therapy per the approved product monograph
* Able to continue methotrexate therapy per the approved product monograph and have received a dose of at least 15 mg/wk (or 10 mg/wk in the case of documented intolerance to higher doses) for at least 12 weeks and this dose has been stable at least 4 weeks before the baseline visit
* The patient or legally acceptable representative must provide written informed consent for participation in the study before any study specific procedures are performed

Exclusion Criteria:

* Patients who have a positive purified protein derivative (PPD) skin test and who do not have a documented course of anti-tuberculosis therapy. Patients with a positive PPD skin test (equal to or greater than 5 mm), a negative chest x-ray at screening which should be repeated if indicated during of the study, at low risk based on exposure and travel and have initiated a course of anti-tuberculosis therapy of which at least 8 weeks have been completed would be eligible for the study. The full course of anti-tuberculosis therapy must be completed
* Patients who have previously received infliximab or adalimumab
* Active infections within 2 weeks of the baseline visit or during the study period
* Any history of human immunodeficiency (HIV) infection, untreated tuberculosis, multiple sclerosis, congestive heart failure, hepatitis B, hepatitis C, cytopenia, prior or current use of cyclophosphamide or malignancy (other than basal cell carcinoma or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix) in the past 5 years
* Women who are pregnant or lactating or of childbearing potential who are not using adequate contraception
* Receipt of any investigational therapy within 4 weeks of the initiation of study medication or during the study period
* Presence of any significant and uncontrolled medical condition, which in the investigator's opinion precludes the use of etanercept, as outlined in the product monograph
* Participants not available for follow-up assessment or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- Canada (23):
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Quispamsis, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Sydney, Nova Scotia
  - Research Site, Bowmanville, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Saint-Eustache, Quebec
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Pope JE, Haraoui B, Thorne JC, Vieira A, Poulin-Costello M, Keystone EC. The Canadian methotrexate and etanercept outcome study: a randomised trial of discontinuing versus continuing methotrexate after 6 months of etanercept and methotrexate therapy in rheumatoid arthritis. Ann Rheum Dis. 2014 Dec;73(12):2144-51. doi: 10.1136/annrheumdis-2013-203684. Epub 2013 Aug 26. PMID 23979914
- [Derived] Keystone EC, Pope JE, Thorne JC, Poulin-Costello M, Phan-Chronis K, Vieira A, Haraoui B; CAMEO Investigators. Two-year radiographic and clinical outcomes from the Canadian Methotrexate and Etanercept Outcome study in patients with rheumatoid arthritis. Rheumatology (Oxford). 2016 Feb;55(2):327-34. doi: 10.1093/rheumatology/kev338. Epub 2015 Sep 11. PMID 26361879
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled 28 June 2008 and last patient was enrolled 07 November 2010.
Pre-assignment Details: A total of 258 participants were enrolled, of whom 205 were randomized after 6 months and 53 were not randomized.
Groups:
- Non-randomized: Enrolled participants received treatment with 50 mg/week subcutaneous etanercept added to existing methotrexate therapy of at least 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses) but discontinued prior to completing this 6 months of treatment.
- Etanercept Alone: After six months of treatment with 50 mg/week subcutaneous etanercept added to existing methotrexate therapy of at least 15 mg/week (or 10 mg/week in case of documented intolerance to higher doses) participants were randomized to discontinue methotrexate (tapered over 6 weeks) and continue etanercept alone for an additional 18 months.
Period: Overall Study
Arm/Group | Non-randomized | Etanercept Alone | Etanercept + Methotrexate
Started | 53 | 98 | 107
Completed | 0 | 50 | 75
Not Completed | 53 | 48 | 32
Not completed — Ineligibility determined | 6 | 0 | 0
Not completed — Protocol deviation | 3 | 2 | 1
Not completed — Non-compliance | 2 | 1 | 2
Not completed — Withdrawal by Subject | 5 | 2 | 2
Not completed — Disease progression | 21 | 31 | 13
Not completed — Requirement for alternative therapy | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Other | 0 | 2 | 3
Not completed — Adverse Event | 14 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-randomized | Etanercept Alone | Etanercept + Methotrexate | Total
Number analyzed (Participants) | 53 | 98 | 107 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (13.4) | 54.3 (11.9) | 54.4 (12.7) | 54.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 72 | 84 | 197
  Male | 12 | 26 | 23 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 47 | 96 | 103 | 246
  Black or African American | 2 | 1 | 0 | 3
  Hispanic or Latino | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 3 | 3
  Aborigine | 1 | 0 | 0 | 1
  Other | 1 | 1 | 0 | 2
Duration of rheumatoid arthritis [Number; unit: participants]
  < 2 years | 11 | 23 | 23 | 57
  >= 2 years | 42 | 75 | 84 | 201
Reimbursement type [Number; unit: participants]
  Private | 23 | 48 | 55 | 126
  Public | 16 | 33 | 37 | 86
  Combination/Other | 14 | 17 | 15 | 46
Disease Activity Score (DAS28-ESR) [Number; unit: participants] — The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • Erythrocyte sedimentation rate (ESR); • Patient's global assessment of disease activity measured on a 100 mm visual analog scale. The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity.
  participants
    <= 5.1 | 20 | 43 | 41 | 104
    > 5.1 | 33 | 55 | 66 | 154

OUTCOME MEASURES:

1. Primary Outcome: Change From Month 6 to Month 12 in Disease Activity Sscore 28 (DAS28)
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • Erythrocyte sedimentation rate (ESR); • Patient's global assessment of disease activity measured on a 100 mm visual analog scale. The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. In this study, the mean change in DAS28 scores from Month 6 to Month 12 was multiplied by a factor of -1, such that a negative change in DAS28 indicates worsening in disease activity.
Time Frame: Month 6 (randomization) and Month 12
Population: The per protocol population defined as all randomized participants with DAS28 measurements both at the 6- and 12-month visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 73 | 88
scores on a scale | -0.39 (0.11) | 0.02 (1.26)
Statistical Analysis 1: Comparison: Etanercept Alone vs Etanercept + Methotrexate; Test type: Non-Inferiority or Equivalence — If the lower bound of the one-sided 95% confidence interval (CI), defined below, exceeded the noninferiority margin of -0.6, then noninferiority was to be concluded; Mean Difference = -0.41, 95% CI 2-sided [-0.75 to -0.06] — The 95% CI was calculated using the mean square error from an analysis of variance (ANOVA) fitted with effects for treatment and covariates of duration of disease, type of reimbursement, and 6 month DAS28

2. Secondary Outcome: Disease Activity Score (DAS) 28 Response
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • Erythrocyte sedimentation rate (ESR); • Patient's global assessment of disease activity measured on a 100 mm visual analog scale. The DAS28 score ranges from zero to ten. Remission is defined by a DAS28 score less than 2.6. Low disease activity is defined by a DAS28 score less than or equal to 3.2. Moderate is defined as a DAS28 higher than 3.2 but lower than or equal to 5.1. DAS28 above 5.1 indicates high disease activity. End of study is Month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat population (all randomized participants); Last observation carried forward (LOCF) imputation was used. At Month 6 data were available for 95 and 105 participants in each treatment group respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
Percentage of participants
  Month 6: Remission | 30.5 [21.3 to 39.8] | 25.7 [17.4 to 34.1]
  Month 6: Low | 16.8 [9.3 to 24.4] | 19.0 [11.5 to 26.6]
  Month 6: Moderate | 41.1 [31.2 to 50.9] | 41.9 [32.5 to 51.3]
  Month 6: High | 11.6 [5.1 to 18.0] | 13.3 [6.8 to 19.8]
  Month 12: Remission | 19.4 [11.6 to 27.2] | 23.4 [15.3 to 31.4]
  Month 12: Low | 10.2 [4.2 to 16.2] | 19.6 [12.1 to 27.2]
  Month 12: Moderate | 49.0 [39.1 to 58.9] | 44.9 [35.4 to 54.3]
  Month 12: High | 21.4 [13.3 to 29.6] | 12.1 [6.0 to 18.3]
  Month 18: Remission | 21.4 [13.3 to 29.6] | 32.7 [23.8 to 41.6]
  Month 18: Low | 12.2 [5.8 to 18.7] | 19.6 [12.1 to 27.2]
  Month 18: Moderate | 41.8 [32.1 to 51.6] | 34.6 [25.6 to 43.6]
  Month 18: High | 24.5 [16.0 to 33.0] | 13.1 [6.7 to 19.5]
  End of Study: Remission | 21.4 [13.3 to 29.6] | 29.9 [21.2 to 38.6]
  End of Study: Low | 8.2 [2.7 to 13.6] | 14.0 [7.4 to 20.6]
  End of Study: Moderate | 45.9 [36.1 to 55.8] | 39.3 [30.0 to 48.5]
  End of Study: High | 24.5 [16.0 to 33.0] | 16.8 [9.7 to 23.9]

3. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28)
Description: The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • Erythrocyte sedimentation rate (ESR); • Patient's global assessment of disease activity measured on a 100 mm visual analog scale. The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. In this study, the mean changes in DAS28 scores from Baseline were multiplied by a factor of -1, such that a negative change in DAS28 indicates worsening in disease activity. End of study is Month 24 or early termination.
Time Frame: Baseline and Month 6, 12, 18 and 24
Population: Intent to treat; LOCF. The number of participants with available data at Month 6 was 95 and 105 in each treatment group respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
scores on a scale
  Change from Baseline to Month 6 | 1.97 (1.23) | 1.97 (1.51)
  Change from Baseline to Month 12 | 1.43 (1.27) | 1.91 (1.61)
  Change from Baseline to Month 18 | 1.35 (1.30) | 2.01 (1.59)
  Change from Baseline to End of Study | 1.37 (1.32) | 1.86 (1.71)

4. Secondary Outcome: Drug Persistence
Description: Drug persistence is defined as the percentage of participants receiving etanercept at 6, 12, 18, and 24 months.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to Treat Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
percentage of participants
  Month 6 | 100 | 100
  Month 12 | 93.2 | 87.6
  Month 18 | 81.9 | 78.8
  Month 24 | 51.4 | 69.5

5. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS)
Description: The modified Total Sharp Score (mTSS) is a measure of change in joint health. X-rays of hands and feet were scored in a blinded manner by an independent reader. Joints were scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (bony ankylosis or complete luxation). Erosion scores and narrowing scores were added to obtain the total mTSS score, ranging from 0 (normal) to 448 (maximal disease). An increase in mTSS from Baseline (represented by a positive change from Baseline score) indicates disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease (negative change from Baseline score) represents improvement. End of study is Month 24 or early termination.
Time Frame: Baseline, Month 12 and Month 24
Population: Radiographic Analysis Set - All randomized participants with a baseline and at least 1 post baseline radiographic assessment. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 94 | 104
scores on a scale
  Change from Baseline to Month 12 (n=89, 102) | 0.3 (1.9) | 0.1 (1.2)
  Change from Baseline to End of Study (n=94, 104) | 0.4 (1.9) | 0.0 (1.4)

6. Secondary Outcome: Change From Baseline in Joint Erosion Score
Description: X-rays of hands and feet were read centrally and in a blinded manner. Sixteen joints on each hand/wrist and 6 joints on each foot were scored for erosions on a scale of 0 to 5 (or for the feet from 0 to 10, with each side of the joint independently scored from 0 to 5) according to the following: One point is scored if erosions are discrete, rising to 2, 3, 4, or 5 depending on the amount of surface area affected (complete collapse of the bone is scored as 5). Scores were summed to calculate the total erosion score, which ranges from 0 (no erosion) to 280 (worst). A large increase in erosion score is indicative of worsening, whereas a small change or no change is indicative of inhibition of joint erosion. End of study is Month 24 or early termination.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 94 | 104
scores on a scale
  Change from Baseline to Month 12 (n=89, 102) | 0.0 (0.6) | 0.0 (0.6)
  Change from Baseline to End of Study (n=94, 104) | 0.1 (0.6) | 0.0 (0.7)

7. Secondary Outcome: Change From Baseline in Joint Space Narrowing
Description: X-rays of hands and feet were read centrally and in a blinded manner. Joint space narrowing (JSN) scores were recorded for each hand/wrist (15 joints) and each foot (6 joints) on a 5-point scale scored as follows:
  0 = normal; 1 = focal or doubtful; 2 = generalised, less than 50% of the original joint space; 3 = generalised, more than 50% of the original joint space or subluxation; 4 = bony ankylosis or complete luxation. The scores were summed to calculate the total JSN score ranging from 0 to 168 (worst). A large increase in joint narrowing score is indicative of worsening, whereas a small change or no change is indicative of inhibition of JSN.
  End of study is Month 24 or early termination.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 94 | 104
scores on a scale
  Change from Baseline to Month 12 (n=89, 102) | 0.2 (1.5) | 0.1 (0.9)
  Change from Baseline to End of Study (n=94, 104) | 0.3 (1.5) | -0.0 (1.0)

8. Secondary Outcome: Change From Month 6 in Health Assessment Questionnaire Disability Index (HAQ DI)
Description: The HAQ disability index is a patient-reported questionnaire specific for rheumatoid arthritis that addresses health-related quality of life. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants choose from four response categories, ranging from 'without any difficulty' (score=0) to 'unable to do' (score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A negative change score indicates an improvement. End of study is Month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat analysis set; LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
scores on a scale
  Change from Month 6 to Month 12 | 0.148 (0.354) | 0.026 (0.430)
  Change from Month 6 to Month 18 | 0.179 (0.452) | -0.004 (0.485)
  Change from Month 6 to End of Study | 0.198 (0.448) | 0.016 (0.539)

9. Secondary Outcome: Change From Month 6 in Health Assessment Questionnaire Pain Visual Analog Scale (VAS)
Description: The HAQ pain visual analog scale (VAS) is a measure of pain on a continuous 100 point scale. Participants were asked to indicate how much pain they had in the past week as a result of their illness on a horizontal line from 0 (no pain) to 100 (severe pain). End of study is Month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat analysis set with available data; LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 106
scores on a scale
  Change from month 6 to month 12 | 7.3 (21.3) | 2.4 (23.8)
  Change from month 6 to month 18 | 8.0 (25.6) | 1.8 (24.4)
  Change from month 6 to end of study | 8.7 (26.1) | 5.1 (27.3)

10. Secondary Outcome: Change From Month 6 in Short Form 36 Health Survey (SF-36)
Description: The SF-36 assesses the general quality of life (QOL) of participants by evaluating the domains of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The questionnaire consists of 36 questions that are completed by the participant.
  The SF-36 is split into two major components: physical health and mental health. Under physical health are the following four domains: physical health, bodily pain, physical functioning and physical role limitations. Under the mental health domain there are four domains; mental health, vitality, social functioning, and emotional role limitation. The individual domain scores are aggregated to derive a physical-component summary score and a mental-component summary score which range from 0 to 100, with higher scores indicating a better level of functioning.
  End of study is month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat analysis set with available SF-36 data at month 6; LOCF
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 106
scores on a scale
  Physical Component: Change at Month 12 | -1.74 (8.87) | -0.30 (7.40)
  Physical Component: Change at Month 18 | -3.28 (9.40) | -0.10 (8.61)
  Physical Component: Change at End of Study | -3.08 (8.95) | -0.75 (9.42)
  Mental Health Component: Change at 12 Months | -1.16 (10.29) | -1.27 (9.40)
  Mental Health Component: Change at 18 Months | -0.30 (9.40) | -0.92 (10.34)
  Mental Health Component: Change at End of Study | -1.30 (10.47) | 0.08 (10.70)

11. Secondary Outcome: Change From Month 6 in Work Productivity and Activity Impairment (WPAI)
Description: This 6-item assessment measures productivity losses during the past 7 days and includes measures on work time missed due to health, impairment while working due to health (the participant's assessment of the degree to which health affected their productivity while working), overall work impairment due to health (takes into account both hours missed due to health and the participant's assessment of the degree to which health affected their productivity while working) and activity impairment due to health (the degree in which health problems affected their ability to do regular daily activities). Scores for each measure are expressed from 0 to 100 with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. For each measure change from Month 6 is reported; a negative change score indicates improvement. End of study is month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat analysis set with available data; Work time missed and work impairment scores are only calculated for participants who were employed at the time. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
scores on a scale
  Work Time Missed: Month 12 (n=45, 44) | -4.2 (19.3) | -0.3 (15.0)
  Work Time Missed: Month 18 (n=42, 43) | -5.5 (20.2) | 0.9 (17.5)
  Work Time Missed: End of Study (n=42, 44) | -3.8 (23.3) | -0.1 (15.6)
  Work Impairment: Month 12 (n=43, 46) | 5.8 (15.0) | -1.3 (19.6)
  Work Impairment: Month 18 (n=40, 45) | 7.3 (24.2) | -1.3 (21.8)
  Work Impairment: End of Study (n=40, 46) | 10.5 (22.2) | -1.7 (24.1)
  Overall Work Impairment: Month 12 (n=43, 44) | 3.4 (16.8) | -0.7 (20.1)
  Overall Work Impairment: Month 18 (n=40, 43) | 4.3 (26.0) | -2.7 (24.2)
  Overall Work Impairment: End of Study (n=40, 44) | 8.2 (26.4) | -1.7 (25.0)
  Activity Impairment: Month 12 (n=98, 107) | 6.7 (21.2) | 4.3 (22.7)
  Activity Impairment: Month 18 (n=98, 107) | 7.4 (25.8) | 0.7 (25.3)
  Activity Impairment: End of Study (n=98, 107) | 9.1 (27.0) | 1.8 (27.4)

12. Secondary Outcome: Change From Month 6 in Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The Treatment Satisfaction Questionnaire for Medication is a 14-item self-administered questionnaire which measures patients' experiences with their medication on four dimensions: effectiveness, side effects, convenience and global satisfaction. Optional responses are: Extremely Dissatisfied (1), Very Dissatisfied (2), Dissatisfied (3), Somewhat Satisfied (4), Satisfied (5), Very Satisfied (6), and Extremely Satisfied (7). For each dimension, responses are added and transformed to a scale from 0 - 100, where higher scores indicate greater satisfaction. Change from Month 6 is reported for each dimension; a positive change score indicates improvement. End of study is Month 24 or early termination.
Time Frame: Month 6, 12, 18 and 24
Population: Intent to treat analysis set with available data; LOCF. n indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
scores on a scale
  Effectiveness: Month 12 (n=98, 107) | -5.0 (27.3) | -1.2 (30.0)
  Effectiveness: Month 18 (n=98, 107) | -7.4 (25.2) | -1.1 (29.4)
  Effectiveness: End of Study (n=98, 107) | -5.0 (25.6) | -1.5 (29.7)
  Side Effects: Month 12 (n= 97, 106) | 2.5 (21.4) | 0.6 (19.0)
  Side Effects: Month 18 (n=97, 106) | -0.5 (24.8) | 0.9 (17.9)
  Side Effects: End of Study (n=97, 106) | 0.6 (24.7) | 1.2 (19.4)
  Convenience: Month 12 (n=97, 107) | 0.6 (16.5) | 0.9 (14.3)
  Convenience: Month 18 (n=97, 107) | 0.9 (15.6) | -0.8 (15.1)
  Convenience: End of Study (n=97, 107) | 2.0 (15.0) | -0.6 (15.3)
  Global Satisfaction: Month 12 (n=97, 107) | -1.3 (19.4) | 1.2 (17.3)
  Global Satisfaction: Month 18 (n=97, 107) | -6.3 (24.0) | -1.5 (20.0)
  Global Satisfaction: End of Study (n=97, 107) | -5.4 (23.7) | -1.3 (20.9)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event (SAE) is defined by regulatory authorities as one that: • is fatal • is life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • other significant medical hazard.
Time Frame: 25 months
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Etanercept Alone | Etanercept + Methotrexate
Number analyzed (Participants) | 98 | 107
participants
  Any adverse event | 86 | 92
  Serious adverse event | 11 | 17
  AEs leading to withdrawal from study drug | 9 | 6

ADVERSE EVENTS:
Time Frame: 25 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Non-randomized | Etanercept Alone | Etanercept + Methotrexate
Serious Adverse Events (participants affected / at risk) | 7/53 | 11/98 | 17/107
Other Adverse Events (participants affected / at risk) | 18/53 | 56/98 | 73/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized (N=53) | Etanercept Alone (N=98) | Etanercept + Methotrexate (N=107)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 2
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized (N=53) | Etanercept Alone (N=98) | Etanercept + Methotrexate (N=107)
Nausea (Gastrointestinal disorders) | 3 | 2 | 6
Fatigue (General disorders) | 1 | 3 | 6
Injection site reaction (General disorders) | 2 | 6 | 7
Bronchitis (Infections and infestations) | 0 | 5 | 7
Influenza (Infections and infestations) | 0 | 7 | 5
Nasopharyngitis (Infections and infestations) | 1 | 10 | 12
Pneumonia (Infections and infestations) | 1 | 1 | 9
Sinusitis (Infections and infestations) | 1 | 8 | 11
Upper respiratory tract infection (Infections and infestations) | 2 | 13 | 19
Urinary tract infection (Infections and infestations) | 4 | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 5 | 10
Headache (Nervous system disorders) | 5 | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.